CLINICAL TRIAL: NCT05562011
Title: A Pilot Feasibility Study of an Ambulatory Multi-Vital Signs Monitor in Perioperative Patients
Brief Title: Feasibility of a New Ambulatory Multi-vital Signs Monitor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: feasibility of device use
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB00073729
Record Dates: First submitted 2022-06-03; First posted 2022-09-30 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-09

CONDITIONS: Perioperative/Postoperative Complications
Keywords: Caretaker; wrist monitor; vital signs
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Caretaker device placement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Caretaker Device (Experimental): participants will undergo active CareTaker monitoring for 24-48 hours
  Interventions: Device: Caretaker Device placement

INTERVENTIONS:
Device: Caretaker Device placement — a continuous non-invasive blood pressure and vital signs monitor that is worn on the wrist

SUMMARY:
The purpose of this research is evaluate vital signs (VS), which include non-invasive blood pressure, pulse rate, respiratory rate and Oxygen Saturation (SpO2) using a portable wrist monitoring device called a Caretaker. This device has been cleared by the Food and Drug Administration (FDA) for use and allows the study team to check vital signs in a participant's normal setting.

Participation in this study will involve wearing this portable device at 2 different time points:

1. for up to 24 hours immediately during and after the participant's preoperative visit to obtain baseline vital signs during normal activity and during sleep and
2. after surgery up to 24 hours while participant recovers prior to discharge from the hospital

DETAILED DESCRIPTION:
Anesthesiologists and surgeons examine vital signs such as heart rate (HR), respiratory rate (RR), oxygen saturation (SaO2) and blood pressure (BP) in an effort to detect extremes of altered VS and remediate these alterations prior to surgery and anesthesia. In most preoperative clinics, however, these VS are measured once and no further assessments are made until they arrive for their surgery. Patients with cardiac and pulmonary disease, however, can have highly variable VS.

The Caretaker device is a wrist device designed to measure relatively continuous VS over a period up to 24 hours. The device is accompanied by a finger cuff that measure pulse and respiratory rate, along with a non-invasive blood pressure detector and pulse oximeter. In an effort to detect VS that may not be recognized with the usual one-time measurement in the clinic, the study team plans to monitor ambulatory preoperative VS in patients who meet the study criteria, for up to 16-24 hours preoperatively. They will then return their device on the day of surgery.

Postoperatively, the study team will place a CareTaker device once again and measure these same VS in the same patients for up to 24 hours prior to discharge.

ELIGIBILITY:
* Inclusion Criteria

  * Age>18 years
  * Scheduled for surgery from an outpatient setting and scheduled for a pre-admission PAC appointment
  * Risk stratification placing them in the top 25th percentile using our internally-validated PAC Risk Score.
* Exclusion Criteria

  * Surgery on the day of admission (same-day surgery)
  * Any upper extremity surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Harwood, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Caretaker Device: participants will undergo active CarTaker monitoring for 24-48 hours
Period: Overall Study
Arm/Group | Caretaker Device
Started | 61
Completed | 39
Not Completed | 22
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Could not co-enroll with other research study--device could not be placed postop | 1
Not completed — Device not placed postop due to patient being discharged home after surgery (not staying overnight) | 4
Not completed — Device malfunction | 13

BASELINE CHARACTERISTICS:
Groups:
- Caretaker Device Placement: Caretaker Device placement: placement of the Caretaker device at preanesthesia visit and again postoperatively
Arm/Group | Caretaker Device Placement
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 31
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Preoperative Caretaker Monitor Placement Success
Description: Number of participants who had the presence of (data existing for at least 70% of 5-minute time periods) for all of the vital signs of interest together--heart rate (HR), blood pressure (BP), respiratory rate (RR), arterial oxygen saturation (SaO2) after placement of the device on the subject's wrist and hand.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
Participants | 39

2. Primary Outcome: Ease of Use Determined by Number of Participants With Sleep or Activities of Daily Living (ADLs) Interference
Description: Participants' description of ease of use (interfered with Activities of Daily Living (ADLs) or sleep) in Yes/No format. Data will be collected to demonstrate percent of patients who answered "Yes" to Sleep or ADL interference. Free text will also be recorded for qualitative purposes. Shows Caretaker Feasibility.
Time Frame: Pre-Op Hour 24
Measure: Count of Participants; unit: Participants
Groups:
- Caretaker Device: Caretaker Device participants will undergo active CareTaker monitoring for 24-48 hours
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
Participants | 16

3. Primary Outcome: Postoperative Caretaker Healthcare Provider (HCP) Usability
Description: Using postoperative nurse verbal feedback on usability of the Caretaker monitor on subjects scheduled for surgery during the perioperative period. Percent of nurses who answer yes to the question: Did you have any difficulty using the Caretaker monitor?
Time Frame: Post-Op Hour 24
Population: Data not collected
Arm/Group | Caretaker Device
Number analyzed (Participants) | 0

4. Primary Outcome: Caretaker Data Capture Rate
Description: Number of participants with no missing values expressed
Time Frame: Pre-Op Hour 24
Population: data not collected
Arm/Group | Caretaker Device
Number analyzed (Participants) | 0

5. Primary Outcome: Caretaker Data Capture Rate
Description: Number of participants with no missing values expressed
Time Frame: Intraoperative; from the time the Operating Room monitors are placed on the patient until they come off at the end of the case, an average of 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
Participants | 39

6. Primary Outcome: Caretaker Data Capture Rate
Description: Number of participants with no missing values expressed
Time Frame: Post-Op Hour 24
Population: data not collected
Arm/Group | Caretaker Device
Number analyzed (Participants) | 0

7. Primary Outcome: Monitor Return Rate
Description: Percent of monitors returned to our research technicians
Time Frame: Baseline through Pre-Op Hour 24
Measure: Count of Participants; unit: Participants
Arm/Group | Caretaker Device
Number analyzed (Participants) | 61
Participants | 61

8. Secondary Outcome: Heart Rate
Time Frame: Pre-Op hour 24, Post-Op Hour 24
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
beats per minute
  Pre-Op Hour 24 | 94 (19)
  Post-Op Hour 24 | 87 (15)

9. Secondary Outcome: Heart Rate--percent of Time Parameters
Description: Percentage of time heart rate is <60 bpm or >90 bpm
Time Frame: Pre-Op Hour 24, Post-Op Hour 24
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
percentage of time
  Pre-Op Hour 24 | 55 (3)
  Post-Op Hour 24 | 40 (4)

10. Secondary Outcome: Respiratory Rate
Time Frame: Pre-Op hour 24, Post-Op Hour 24
Measure: Mean (Standard Deviation); unit: respirations per minute
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
respirations per minute
  Pre-Op Hour 24 | 17 (4)
  Post-Op Hour 24 | 17 (4)

11. Secondary Outcome: Respiratory Rate--Percent of Time Parameters
Description: Percent of time respirations are <8 rpm or >20 rpm
Time Frame: Pre-Op hour 24, Post-Op Hour 24
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
percentage of time
  Pre-Op Hour 24 | 21.6 (3.8)
  Post-Op Hour 24 | 15.9 (3.5)

12. Secondary Outcome: Arterial Oxygen Saturation (SaO2)
Description: oxygen saturation level as detected by the pulse oximeter
Time Frame: Post-Op Hour 24
Population: data not collected
Arm/Group | Caretaker Device
Number analyzed (Participants) | 0

13. Secondary Outcome: SaO2--Percent of Time
Description: Percentage of time SaO2 is between 95-100%
Time Frame: Pre-Op Hour 24, Post-Op Hour 24
Population: data not collected for either time point
Arm/Group | Caretaker Device
Number analyzed (Participants) | 0

14. Secondary Outcome: Non-Invasive Systolic Blood Pressure (SBP)
Time Frame: Pre-Op Hour 24, Post-Op Hour 24
Measure: Mean (Standard Deviation); unit: units of millimeters of mercury (mmHg)
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
units of millimeters of mercury (mmHg)
  Pre-Op Hour 24 | 119 (22)
  Post-Op Hour 24 | 134 (24)

15. Secondary Outcome: Non-Invasive Mean Arterial Blood Pressure (MBP)
Time Frame: Pre-Op Hour 24, Post-Op Hour 24
Measure: Mean (Standard Deviation); unit: mm of Hg
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
mm of Hg
  Pre-Op Hour 24 | 82 (18)
  Post-Op Hour 24 | 97 (21)

16. Secondary Outcome: Non-Invasive Diastolic Blood Pressure (DBP)
Time Frame: Pre-Op Hour 24, Post-Op Hour 24
Measure: Mean (Standard Deviation); unit: mm of Hg
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
mm of Hg
  Pre-Op Hour 24 | 58 (16)
  Post-Op Hour 24 | 68 (16)

17. Secondary Outcome: Non-Invasive Blood Pressure--MBP Percent of Time Parameters
Description: Percent time MBP is <60 mmHg and/or >90 mmHg
Time Frame: Pre-Op Hour 24, Post-Op Hour 24
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
percentage of time
  Pre-Op Hour 24 | 37 (4)
  Post-Op Hour 24 | 67 (1)

18. Secondary Outcome: Mortality Rate
Description: Percent declared dead
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Caretaker Device
Number analyzed (Participants) | 61
Participants | 0

19. Secondary Outcome: Average Length of Hospital Stay
Description: Number of days from hospital admission to discharge
Time Frame: Up to Postoperative Day 30
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
number of days | 3.5 (4.3)

20. Secondary Outcome: ICU Transfer Rate
Description: Percent of study participants transferred to an ICU during their hospital stay
Time Frame: Up to Postoperative Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
Participants | 10

21. Secondary Outcome: Number of Rapid Response Team Calls
Description: Number of calls made to the hospital's "Rapid Response Team" (RRT) during subjects' hospital stay. The RRT is called by nurses if the patient is experiencing stroke-like symptoms, chest pain refractory to medical treatment, or vital signs (HR, RR, BP, SaO2) meeting a pre-defined out of range value.
Time Frame: During hospitalization up to Postoperative Day 30
Measure: Number; unit: calls
Arm/Group | Caretaker Device
Number analyzed (Participants) | 39
calls | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Caretaker Device
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT05562011/Prot_SAP_002.pdf
  • Informed Consent Form (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT05562011/ICF_001.pdf